CLINICAL TRIAL: NCT01627041
Title: Randomized Phase II Study of Epigenetic Priming Using Decitabine With Induction Chemotherapy in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Decitabine, Cytarabine, and Daunorubicin Hydrochloride in Treating Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01959; NCI-2012-01959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1106011736; CDR0000712322; 1106011736 (Other: NYP/Weill Cornell Medical Center); 8854 (Other: CTEP); N01CM00070 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Basophilic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With t(9;11)(p21.3;q23.3); MLLT3-KMT2A; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Basophilic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute | interventions — Cytarabine; Daunorubicin; Decitabine; Injections

ARMS (2):
- Arm I (daunorubicin hydrochloride, cytarabine) (Experimental): Patients receive induction chemotherapy comprising daunorubicin hydrochloride IV daily on days 1-3 and cytarabine IV continuously on days 1-7 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR after the first induction-chemotherapy course receive a second identical induction course.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (decitabine, daunorubicin hydrochloride, cytarabine) (Experimental): Patients receive decitabine IV over 1 hour on days -5 to -1. Patients then receive induction chemotherapy as in arm I in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR after the first induction-chemotherapy course receive a second identical induction course.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Arm II (decitabine, daunorubicin hydrochloride, cytarabine)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial studies how well decitabine works when given together with daunorubicin hydrochloride and cytarabine in treating patients with acute myeloid leukemia. Drugs used in chemotherapy, such as decitabine, daunorubicin hydrochloride, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Decitabine may help daunorubicin hydrochloride and cytarabine kill more cancer cells by making them more sensitive to the drugs. It is not yet known whether low-dose decitabine is more effective than high-dose decitabine when giving together with daunorubicin hydrochloride and cytarabine in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. To "Pick a Winner" by deciding whether further development of epigenetic priming with decitabine prior to standard "7+3" induction chemotherapy should be pursued.

Secondary I. To determine whether epigenetic priming with decitabine prior to standard cytarabine and daunorubicin hydrochloride "7+3" induction chemotherapy has sufficient efficacy to warrant further development as assessed by an overall CR1 rate ≥ 50%.

II. To establish the safety and expected toxicities of decitabine when used as priming for cytarabine and daunorubicin hydrochloride "7+3" induction chemotherapy in acute myeloid leukemia (AML).

III. To assess the pharmacodynamics of deoxyribonucleic acid (DNA) hypomethylation when decitabine is administered as a short infusion.

IV. To investigate, in selected cases, the molecular and cellular consequences of decitabine-induced hypomethylation by assessing the effects of decitabine-mediated hypomethylation on transcriptional patterns in AML cells, and by determining the effect of hypomethylation on the differentiation and/or apoptosis of leukemic blasts. (exploratory) V. To identify biomolecular correlates of treatment response (biomarkers) to induction chemotherapy in AML based upon the epigenetic pattern of DNA methylation in AML specimens obtained prior to treatment. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to age (less than 50 years vs 50-65 years), white blood cell count (≤ 30 K/mL vs greater than 30 K/mL), cytogenetic risk group (intermediate vs adverse risk), and antecedent hematological condition preceding the diagnosis of acute myeloid leukemia (yes vs no). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive induction chemotherapy comprising daunorubicin hydrochloride intravenously (IV) daily on days 1-3 and cytarabine IV continuously on days 1-7 in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a complete remission (CR) after the first induction-chemotherapy course receive a second identical induction course.

Arm II: Patients receive decitabine IV over 1 hour on days -5 to -1. Patients then receive induction chemotherapy as in arm I in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR after the first induction-chemotherapy course receive a second identical induction course.

Patients undergo blood, bone marrow, and oral mucosa cells sample collection at baseline, prior to induction therapy, and after treatment for DNA methylation studies and pharmacodynamic studies.

After completion of study treatment, patients are followed up for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) as defined by the World Health Organization
* Molecular AML-risk group is less-than-favorable as defined by any of the following criteria:

  * The absence of good-risk karyotype t(8;21), inv(16), t(16;16), or t(15;17)identified by metaphase karyotype
  * The absence of t(8;21), inv(16), t(16;16), or t(15;17) identified by fluorescent in situ hybridization(FISH)
  * The absence of the corresponding fusion transcripts, AML1-eight-twenty-one corepressor (ETO), core-binding factor, beta subunit (CBFβ)-smooth muscle myosin heavy chain (SMMHC), or progressive multifocal leukoencephalopathy (PML)-retinoic acid receptor alpha (RARa), identified by reverse transcriptase-polymerase chain reaction (RT-PCR)
  * Patient does not have acute promyelocytic leukemia (APL, French-American-British [FAB] M3)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Adequate cardiac function as defined by either of the following:

  * An echocardiogram demonstrating an ejection fraction within normal limits
  * A multi gated acquisition (MUGA) scan demonstrating an ejection fraction within normal limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 times institutional upper limit of normal (ULN)
* Creatinine ≤ 2 mg/dL OR creatinine clearance ≥ 50 mL/min
* Total bilirubin ≤ 2 times ULN

  * Patients with documented diagnosis of Gilbert syndrome resulting in elevated total bilirubin levels will be eligible, provided all other eligibility criteria are met
  * Patients with a total bilirubin of 2-3 mg/dL and direct (conjugated) bilirubin in the normal range will be eligible, provided all other eligibility criteria are met
* Pregnant and nursing subjects may not be enrolled and pregnancy must be avoided; women of child-bearing potential-defined as a sexually active woman who has not undergone hysterectomy and who has had menses any time within the preceding 24 months-must have a negative serum or urine pregnancy test within 7 days prior to registration; women and men of childbearing potential must either commit to continued abstinence from heterosexual intercourse or commit to two acceptable methods of birth control-one highly effective method (e.g., IUD, oral or non-oral hormonal contraceptive, tubal ligation or partner's vasectomy) and one additional effective method (e.g., latex condom, diaphragm or cervical cap) at the same time from the time of screening through final Treatment Response Assessment

  * NOTE: should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the subject should inform their treating phy-sician immediately
  * NOTE: the effects of decitabine on the developing human fetus are unknown but it is a know teratogen in mammals (mice)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy (other than hydroxyurea) or radiation within the 2 weeks prior to planned therapy on this study or ongoing adverse events due to agents administered more than 2 weeks earlier
* Concurrent treatment with other investigational agents is not permitted
* Cumulative lifetime dose of anthracycline chemotherapeutic > 80 mg/m^2
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of decitabine, cytarabine or daunorubicin
* Uncontrolled intercurrent illness considered by the investigator to constitute an unwarranted high risk for investigational drug treatment; examples include, but not limited to the following:

  * Uncontrolled serious infection; or
  * Unstable angina pectoris; or
  * Uncontrolled cardiac arrhythmia; or
  * Active second malignancy requiring treatment; or
  * Symptomatic congestive heart failure
* HIV-positive subjects with a CD4 count < 200 cells/μL are excluded due to the increased risk of lethal infections when treated with marrow-suppressive chemotherapy(87)

  * NOTE: subjects with HIV infection and a CD4 count >= 200 cells/μL are eligible but combination antiretroviral therapy should be held during administration of chemotherapy due to the potential for pharmacokinetic interactions with decita-bine, cytarabine or daunorubicin. Antiretroviral therapy may be resumed 24 hours after completion of the last dose of induction chemotherapy
* Subject has a psychiatric disorder, altered mental status or social situation that would preclude understanding of the informed consent process and/or limit compliance with study requirements
* Subject has an inability or unwillingness, in the opinion of the investigator, to comply with the protocol requirements
* Subjects with central nervous system (CNS) (or leptomeningeal) infiltration by AML may be considered for treatment at the Investigator's discretion and following discussion with the Principle Investigator; all neurologic deficits must be noted prior to enrollment on study
* Subject has circulating blast count > 50,000/μL (subjects may be enrolled if circulating blast count is controlled by hydroxyurea and/or, if clinically indicated, by leukophoresis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR1) | After 1 course of decitabine-primed induction chemotherapy

SECONDARY OUTCOMES:
Complete remission rate (CR1 + CR2) | After up to 2 courses of decitabine-primed induction chemotherapy
Overall survival | Time from entry on study to time of death from any cause, assessed up to 10 years
Relapse-free survival | Time from CR documentation to either AML relapse or death from any cause, assessed up to 10 years
Event-free survival | Time from entry on study until treatment failure (no CR with up to two study induction cycles), AML relapse, or death from any cause, assessed up to 10 years
Time to complete response determined according to the International Working Group (IWG) criterion | Time from entry on study until documentation of CR, up to second course of induction chemotherapy
  95% confidence limits will be provided.
Remission duration | Time from CR documentation to either AML relapse, assessed up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Scandura, Principal Investigator — Weill Medical College of Cornell University
Locations (9):
- United States (9):
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio